CLINICAL TRIAL: NCT01309828
Title: A Randomized, Open-Label, Phase 3 Study to Compare Long-Term Safety and Tolerability of the TAK-491 and Chlorthalidone Fixed-Dose Combination Versus Olmesartan Medoxomil and Hydrochlorothiazide Fixed-Dose Combination in Hypertensive Subjects With Moderate Renal Impairment
Brief Title: Long-Term Safety of Azilsartan Medoxomil and Chlorthalidone Compared to Olmesartan Medoxomil and Hydrochlorothiazide in Participants With Hypertension and Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-491CLD_309; 2010-023098-21 (EudraCT Number); U1111-1119-5131 (Registry Identifier: WHO); NL35552.072.11 (Registry Identifier: CCMO)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-09

CONDITIONS: Safety
Keywords: Renal Insufficiency; Kidney Diseases; Hypertension; Drug Therapy
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Hypertension | interventions — azilsartan medoxomil; Chlorthalidone; Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azilsartan Medoxomil + Chlorthalidone (Experimental): United States and Europe: Azilsartan medoxomil 20 mg plus chlorthalidone 12.5 mg fixed dose combination tablets, titrated up to azilsartan medoxomil 40 mg plus chlorthalidone 25 mg orally, once daily for up to 52 weeks.
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Olmesartan Medoxomil + Hydrochlorothiazide (Active Comparator): United States: Olmesartan medoxomil 20 mg plus hydrochlorothiazide 12.5 mg fixed dose combination tablets, titrated up to olmesartan medoxomil 40 mg plus hydrochlorothiazide 25 mg orally, once daily for up to 52 weeks. Europe: Olmesartan medoxomil 20 mg plus hydrochlorothiazide 12.5 mg fixed dose combination tablets, titrated up to olmesartan medoxomil 20 mg plus hydrochlorothiazide 25 mg orally, once daily for up to 52 weeks.
  Interventions: Drug: Olmesartan medoxomil and hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Fixed-dose combination tablets.
  Other Names: TAK-491CLD
  Arms: Azilsartan Medoxomil + Chlorthalidone
Drug: Olmesartan medoxomil and hydrochlorothiazide — Fixed-dose combination tablets.
  Other Names: Olmesartan medoxomil; Hydrochlorothiazide; Benicar hydrochlorothiazide; Olmetec Plus
  Arms: Olmesartan Medoxomil + Hydrochlorothiazide

SUMMARY:
The purpose of this study is to evaluate long term safety and tolerability of azilsartan medoxomil and chlorthalidone, once daily (QD), compared with olmesartan medoxomil and hydrochlorothiazide in hypertensive participants with moderate renal impairment.

DETAILED DESCRIPTION:
A major component of blood pressure regulation is the renin-angiotensin-aldosterone system (RAAS). Drugs that modulate the RAAS are used commonly worldwide for the treatment of hypertension. TAK-491 (azilsartan medoxomil) is a prodrug of TAK-536 (azilsartan), an angiotensin II receptor blocker (ARB). Azilsartan medoxomil is being evaluated by Takeda to treat participants with essential hypertension.

Chlorthalidone is an orally administered thiazide-like diuretic agent, and long-term outcomes trials show blood pressure reductions associated with chlorthalidone treatment reduce risk of cardiovascular morbidity and mortality.

Hypertensive patients with moderate renal impairment are a relatively more severe and resistant hypertension population, and may benefit from effective fixed-dose combination treatments such as an ARB plus a diuretic for blood pressure control.

Participants will be randomized to receive azilsartan medoxomil and chlorthalidone or olmesartan medoxomil and hydrochlorothiazide for up to 52 weeks to evaluate long term safety of azilsartan medoxomil and chlorthalidone. A titration-to-target blood pressure approach will be used to guide the titration of study medication in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Is treated with 2 or 3 antihypertensive medications and on stable therapy, defined as ≥6 weeks on medication, and has a mean sitting clinic systolic blood pressure ≥135 and ≤160 mm Hg at the Screening Visit and on Day 1.
2. Has an estimated glomerular filtration rate (eGFR) in the range of ≥30 to <60 mL/min/1.73 m^2 (Stage 3 chronic kidney disease) at the Screening Visit.
3. Is a man or woman and aged 18 years or older.
4. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent through 30 days after the last study drug dose.
5. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
6. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
7. Has clinical laboratory test results (clinical chemistry, hematology, and complete urinalysis) that the investigator does not consider to be clinically significant in this moderate renal impaired population.
8. Is willing to discontinue the current antihypertensive medications 2 days prior to randomization.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening or is currently participating in another investigational study.
2. Has been randomized/enrolled in a previous TAK-491 or TAK-491CLD study. NOTE: This criterion does not apply to participants who began participation in another TAK-491 or TAK-491CLD study but were not randomized/enrolled, nor does it apply to participants who participated in observational studies that lacked an intervention or invasive procedure.
3. Is receiving a combination of olmesartan and hydrochlorothiazide at the Screening Visit.
4. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
5. Has a mean clinic diastolic (sitting, trough) >110 mm Hg on Day 1.
6. Has secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
7. Has a recent history (within the last 6 months) of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
8. Has clinically significant cardiac conduction defects (ie, third-degree atrioventricular block, sick sinus syndrome).
9. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
10. Has severe renal dysfunction or disease (based on eGFR <30 mL/min/1.73m^2 at Screening) prior renal transplantation or nephrotic syndrome (defined as a urinary albumin/creatinine ratio >2000 mg/g at Screening).
11. Has known or suspected unilateral or bilateral renal artery stenosis.
12. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those participants with basal cell or stage I squamous cell carcinoma of the skin.)
13. Has poorly-controlled type 1 or 2 diabetes mellitus (glycosylated hemoglobin A [HbA1c] >8.5%) at Screening.
14. Has hypokalemia or hyperkalemia (defined as serum potassium outside of the normal reference range of the central laboratory).
15. Has an alanine aminotransferase or aspartate aminotransferase level of >2.5 times the upper limit of normal, active liver disease, or jaundice.
16. Has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
17. has a history of hypersensitivity or allergies to ARBs or thiazide-type diuretics or other sulfonamide-derived compounds.
18. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within the past 2 years.
19. Is required to take excluded medications.
20. If female, is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (53):
- Bulgaria (5):
  - Kazanlak
  - Pleven
  - Sevlievo
  - Sofia
  - Varna
- Germany (10):
  - Mannheim, Baden-Wurttemberg
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Offenbach, Hesse
  - Rodgau Dudenhofen, Hesse
  - Essen, North Rhine-Westphalia
  - Goch, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Berlin, State of Berlin
- Latvia (6):
  - Daugavpils
  - Kuldīga
  - Limbaži
  - Riga
  - Tukums
  - Ventspils
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Maastricht
  - Venlo
- Poland (5):
  - Grodzisk Mazowiecki
  - Lodz
  - Torun
  - Warsaw
  - Zgierz
- Slovakia (9):
  - Banská Bystrica
  - Bardejov
  - Bratislava
  - Komárno
  - Košice
  - Martin
  - Nitra
  - Ružomberok
  - Svidník
- Ukraine (9):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lutsk
  - Lviv
  - Vinnitsya
  - Vinnytsia

REFERENCES:
- [Derived] Bakris GL, Zhao L, Kupfer S, Juhasz A, Hisada M, Lloyd E, Oparil S. Long-term efficacy and tolerability of azilsartan medoxomil/chlorthalidone vs olmesartan medoxomil/hydrochlorothiazide in chronic kidney disease. J Clin Hypertens (Greenwich). 2018 Apr;20(4):694-702. doi: 10.1111/jch.13230. Epub 2018 Mar 4. PMID 29504252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 46 investigative sites in the United States, Germany, Latvia, Lithuania, Poland, Slovakia, and the Ukraine from 02 March 2011 to 11 October 2012.
Pre-assignment Details: Participants with high blood pressure and moderate renal impairment were enrolled in 1 of 2 once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil + Chlorthalidone: United States and Europe: Azilsartan medoxomil 20 mg plus chlorthalidone 12.5 mg fixed dose combination tablets (TAK-491CLD), titrated up to azilsartan medoxomil 40 mg plus chlorthalidone 25 mg orally, once daily for up to 52 weeks.
- Olmesartan Medoxomil + Hydrochlorothiazide: United States: Olmesartan medoxomil 20 mg plus hydrochlorothiazide 12.5 mg fixed dose combination tablets (OLM/HCTZ), titrated up to olmesartan medoxomil 40 mg plus hydrochlorothiazide 25 mg orally, once daily for up to 52 weeks. Europe: Olmesartan medoxomil 20 mg plus hydrochlorothiazide 12.5 mg fixed dose combination tablets, titrated up to olmesartan medoxomil 20 mg plus hydrochlorothiazide 25 mg orally, once daily for up to 52 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Started | 77 | 76
Completed | 61 | 60
Not Completed | 16 | 16
Not completed — Adverse Event | 10 | 11
Not completed — Voluntary Withdrawal | 5 | 4
Not completed — Major Protocol Deviation | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide | Total
Number analyzed (Participants) | 77 | 76 | 153
Age Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.24) | 68.9 (9.10) | 68.4 (8.66)
Age, Customized [Number; unit: participants]
  <45 years | 0 | 1 | 1
  ≥45 to <65 years | 21 | 18 | 39
  ≥65 to <75 years | 38 | 39 | 77
  ≥75 years | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 31 | 76
  Male | 32 | 45 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57 | 62 | 119
  Black or African American | 18 | 12 | 30
  Asian | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 9 | 19
  Latvia | 4 | 5 | 9
  Lithuania | 5 | 2 | 7
  Poland | 7 | 6 | 13
  Slovakia | 6 | 6 | 12
  Ukraine | 6 | 11 | 17
  United States | 39 | 37 | 76
Weight [Mean (Standard Deviation); unit: kg] | 83.54 (17.894) | 90.14 (21.587) | 86.82 (20.025)
Height [Mean (Standard Deviation); unit: cm] | 165.7 (9.65) | 168.7 (9.48) | 167.2 (9.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.44 (6.226) | 31.57 (6.524) | 31.00 (6.380)
Smoking Classification [Number; unit: participants]
  Never Smoked | 46 | 40 | 86
  Current Smoker | 11 | 11 | 22
  Ex-smoker | 20 | 25 | 45
Diabetes Status [Number; unit: participants]
  Yes | 33 | 32 | 65
  No | 44 | 44 | 88
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 48.25 (10.205) | 47.73 (8.761) | 47.99 (9.487)
Baseline estimated glomerular filtration rate (eGFR) category [Number; unit: participants]
  ≥45 and <60 mL/min/1.73 m^2 | 40 | 39 | 79
  ≥30 and <45 mL/min/1.73 m^2 | 31 | 33 | 64
  ≥60 mL/min/1.73 m^2 | 6 | 4 | 10
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 151.1 (10.30) | 149.0 (7.80) | 150.1 (9.18)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 84.8 (10.31) | 84.7 (9.68) | 84.7 (9.97)
Systolic blood pressure categories [Number; unit: participants]
  <140 mm Hg | 11 | 10 | 21
  ≥140 to <160 mm Hg | 60 | 64 | 124
  ≥160 to <180 mm Hg | 5 | 2 | 7
  ≥180 mm Hg | 1 | 0 | 1
Diastolic blood pressure categories [Number; unit: participants]
  <90 mm Hg | 52 | 50 | 102
  ≥90 mm Hg | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have a causal relationship with this treatment. A serious AE is defined as any untoward medical occurrence that resulted in death, was life threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability or incapacity, led to a congenital anomaly/birth defect or was an important medical event that may have required intervention to prevent any of items above.
Time Frame: From the first dose of open-label study drug until 14 days (or 30 days for a serious adverse event) after the last dose of open- label study drug (up to 56 weeks).
Population: Safety analysis set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: participants
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Number analyzed (Participants) | 77 | 76
participants
  Adverse Events | 68 | 58
  Adverse Events Leading to Discontinuation | 17 | 15
  Serious Adverse Events | 8 | 9
  Serious Adverse Events Leading to Discontinuation | 5 | 4
  Death | 0 | 1

2. Secondary Outcome: Percentage of Participants at Final Visit Who Achieve Target Systolic Blood Pressure <130 mm Hg
Description: Systolic blood pressure is the arithmetic mean of the 3 serial sitting systolic blood pressure measurements. Percentage of participants who achieve a sitting clinic systolic blood pressure response defined as less than 130 mm Hg at Week 52.
Time Frame: Week 52
Population: Full analysis set participants (all randomized participants who received at least 1 dose of open-label study drug) with both Baseline and a post-baseline value; last observation carried forward was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Number analyzed (Participants) | 75 | 74
percentage of participants | 69.3 [57.6 to 79.5] | 78.4 [67.3 to 87.1]

3. Secondary Outcome: Percentage of Participants at Final Visit Who Achieved Target Diastolic Blood Pressure <80 mm Hg
Description: Diastolic blood pressure is the arithmetic mean of the 3 serial sitting diastolic blood pressure measurements. Percentage of participants at Week 52 who achieved a sitting clinic diastolic blood pressure response, defined as less than 80 mm Hg.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Number analyzed (Participants) | 75 | 74
percentage of participants | 80.0 [69.2 to 88.4] | 87.8 [78.2 to 94.3]

4. Secondary Outcome: Percentage of Participants at Final Visit Who Achieved Both a Clinic Systolic and Diastolic Blood Pressure Response
Description: Systolic/diastolic blood pressure is the arithmetic mean of the 3 serial sitting systolic/diastolic blood pressure measurements. Percentage of participants who achieved both a sitting clinic systolic and diastolic blood pressure response, defined as systolic blood pressure less than 130 mm Hg and diastolic blood pressure less than 80 mm Hg at Week 52.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Number analyzed (Participants) | 75 | 74
percentage of participants | 58.7 [46.7 to 69.9] | 73.0 [61.4 to 82.6]

ADVERSE EVENTS:
Time Frame: From the first dose of open-label study drug until 14 days (or 30 days for a serious adverse event) after the last dose of open-label study drug (up to 56 weeks).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil + Chlorthalidone | Olmesartan Medoxomil + Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 8/77 | 9/76
Other Adverse Events (participants affected / at risk) | 52/77 | 41/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil + Chlorthalidone (N=77) | Olmesartan Medoxomil + Hydrochlorothiazide (N=76)
Angina unstable (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Device malfunction (General disorders) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil + Chlorthalidone (N=77) | Olmesartan Medoxomil + Hydrochlorothiazide (N=76)
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 3 | 4
Bronchitis (Infections and infestations) | 4 | 3
Pharygitis (Infections and infestations) | 0 | 4
Blood creatinine increased (Investigations) | 34 | 29
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Dizziness (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 8 | 2
Hypotension (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.